CLINICAL TRIAL: NCT04183920
Title: To Determine the Activity and Mechanisms of Cranberries to Attenuate Skin Photoaging and Improve Skin Health in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201903250
Record Dates: First submitted 2019-11-22; First posted 2019-12-03 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Skin Health

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Participants in this arm will be provided cranberry juice to consume for 42 days in total. After a 10-21-day washout period participants will receive placebo juice for 42 days.
  Interventions: Other: Cranberry juice; Other: Placebo juice
- Group B (Active Comparator): Participants in this arm will be provided placebo juice to consume for 42 days in total. After a 10-21-day washout period participants will receive cranberry juice to consume for 42 days
  Interventions: Other: Cranberry juice; Other: Placebo juice

INTERVENTIONS:
Other: Cranberry juice — cranberry juice cocktail provided by Ocean Spray Cranberries, Inc.
Other: Placebo juice — apple juice added with flavor and colorants provided by Ocean Spray Cranberries, Inc.

SUMMARY:
Previous studies have shown that cranberry phytochemicals scavenge reactive carbonyls. Cranberry polyphenols have been reported to attenuate collagen degradation and inhibit oxidative stress in human cells. We hypothesize that cranberry juice consumption will attenuate skin photoaging and improve skin health in women via alleviate oxidative stress.

DETAILED DESCRIPTION:
One of the causative factors of skin ageing is cumulative oxidative damages due to aerobic metabolism and UV irradiation. Cumulation of reactive oxygen species (ROS) causes collagen glycation and crosslinking which are direct causes of skin ageing. Previous studies have shown that cranberry phytochemicals scavenge reactive carbonyls. Cranberry polyphenols have been reported to attenuate collagen degradation and inhibit oxidative stress in human cells. It is unknown whether cranberry juice consumption could protect against UV -induced erythema and improve overall skin health. Furthermore, if it does have effect, what will be the mechanism? This human intervention study will be conducted to answer these questions. We hypothesize that cranberry juice consumption will attenuate skin photoaging and improve skin health in women via alleviate oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI (18.5-29.9)
* Body weight ≥110 pounds

Exclusion Criteria:

* Skin Cancer
* Smokers and frequent alcohol use
* Pregnancy
* Breast-feeding
* intake of medication that might influence the outcome of the study
* sunbathing or the use of tanning bed
* intake of vitamin/mineral supplements

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline Skin color change after UV irradiation at 28 days | Baseline, 28 days
  Irradiation will be applied to dorsal skin (region not typically exposed to the sun) using an FDA approved UVB phototherapy light and a UV light meter. At each assessment, skin color will be measured before and 24 h after irradiation. Skin color will be evaluated by a colorimeter using the 3-dimensional color system with L-, a-, and b-values. L- and b- values assess lightness and browning effects, respectively. The a-value (red/green-axis) is a measure for reddening (erythema). The Δa-values (a-value 24 h after irradiation minus a-value before irradiation) will compared between baseline through 3 months; decreasing Δa-values indicates a photoprotective effect.
Change from baseline Skin transepidermal water loss | Baseline, 28 days
  Skin transepidermal water loss an will be measured using a Tewameter (CK Electronic GmbH, Germany). This is a handheld probes that allow for quick and easy measurements
Change from baseline SELS parameters | Baseline, 28 days
  SELS (Surface evaluation of the Living Skin) parameters, including smoothness, roughness, scaliness, and wrinkles, will be determined using a Visioscan VC20. This hand-hold device scans a 1 cm x 1 cm skin area (https://www.courage-khazaka.de/en/scientific-products/all-products/imaging/16-wissenschaftliche-produkte/alle-produkte/150-visioscan-e). Visioscan VC20 scanner consists of a camera, a high- resolution video sensor, and a UVA light no hazardous to human skin.
Change in skin microbiome | Baseline, 28 days
  For skin swabbing, a 4x4-cm square on a forearm will be swabbed with a cotton swab soaked in 0.9% sodium chloride with 0.1% Tween-20 in a Z-stroke manner.
Change in baseline skin pH | Baseline, 28 days
  Skin pH will be assessed using a skin pH meter (CK Electronic GmbH, Germany). This is a handheld probes that allow for quick and easy measurements.
Change from baseline hydration | Baseline, 28 days
  Skin hydration will be measured with a Corneometer (CK Electronic GmbH, Germany. This is a handheld probe that allows for quick and easy measurements.
Change in Skin erythema and melanin index | Baseline, 28 days
  Skin erythema and melanin index will be assessed with a Mexameter, (CK Electronic GmbH, Germany). Each of these are handheld probes that allow for quick and easy measurements
Change in skin lipidome | baseline, 28 days
  Stratum corneum layer on forearm skin will be sampled with 16 D-squame® tapes using a standard noninvasive tape stripping technique. This will be sent for lipidomic analysis

SECONDARY OUTCOMES:
Survival rate of human keratinocyte under UV light | 24 hours
  The immortalized human keratinocyte cell line (HaCaT) will be cultured in Dulbecco's Modified Eagle Medium. Cells will be incubated with human serum collected after 2-hour and 4-hour cranberry juice intake or water intake for 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Gu, PhD, Principal Investigator — University of Florida
Locations (1):
- Food Science and human nutrition department at University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramasamy R, Yan SF, Schmidt AM. Receptor for AGE (RAGE): signaling mechanisms in the pathogenesis of diabetes and its complications. Ann N Y Acad Sci. 2011 Dec;1243:88-102. doi: 10.1111/j.1749-6632.2011.06320.x. PMID 22211895
- [Background] Liu H, Liu H, Wang W, Khoo C, Taylor J, Gu L. Cranberry phytochemicals inhibit glycation of human hemoglobin and serum albumin by scavenging reactive carbonyls. Food Funct. 2011 Aug;2(8):475-82. doi: 10.1039/c1fo10087d. Epub 2011 Aug 8. PMID 21826359
- [Background] Heinrich U, Moore CE, De Spirt S, Tronnier H, Stahl W. Green tea polyphenols provide photoprotection, increase microcirculation, and modulate skin properties of women. J Nutr. 2011 Jun;141(6):1202-8. doi: 10.3945/jn.110.136465. Epub 2011 Apr 27. PMID 21525260
- [Background] Heinrich U, Neukam K, Tronnier H, Sies H, Stahl W. Long-term ingestion of high flavanol cocoa provides photoprotection against UV-induced erythema and improves skin condition in women. J Nutr. 2006 Jun;136(6):1565-9. doi: 10.1093/jn/136.6.1565. PMID 16702322